CLINICAL TRIAL: NCT06270108
Title: The Role of Glutamatergic Function in the Pathophysiology of Treatment-resistant Schizophrenia
Acronym: RESTORE
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 22/SS/0040; 299382 (Other: Integrated Research Application System)
Record Dates: First submitted 2024-01-29; First posted 2024-02-21 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Treatment-resistant Schizophrenia; Treatment-responsive Schizophrenia; Healthy Controls
Keywords: schizophrenia; treatment-resistant schizophrenia; glutamate; riluzole
MeSH Terms: conditions — Schizophrenia, Treatment-Resistant; Schizophrenia | interventions — Riluzole

STUDY DESIGN:
Intervention Model Description: This is a basic science study the purpose of which is to to explore the responsivity of glutamate in treatment-resistant schizophrenia to a given challenge (riluzole).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment-resistant schizophrenia patients receiving riluzole (Experimental)
  Interventions: Drug: Riluzole
- Treatment-responsive schizophrenia patients (No Intervention)
- Healthy controls (No Intervention)

INTERVENTIONS:
Drug: Riluzole — 50mg twice daily (100mg total daily) for 56 days.
  Arms: Treatment-resistant schizophrenia patients receiving riluzole

SUMMARY:
The goal of this basic science study is to to explore the responsivity of glutamate in the brain of treatment-resistant schizophrenia patients to the drug riluzole. The main aims of the study are:

To assess the role of glutamate in treatment-resistant schizophrenia using magnetic resonance spectroscopy.

To assess the relationship between glutamate levels and brain structural and functional measures (using: structural MRI; functional MRI (fMRI) and arterial spin labelling (ASL)) at baseline.

To assess the relationship between longitudinal change in glutamate levels and brain structural and functional measures.

To assess the relationship between longitudinal change in glutamate levels and changes in psychopathology.

The researchers will compare the changes with healthy controls and those without treatment-resistant schizophrenia.

ELIGIBILITY:
Inclusion criteria for treatment-resistant schizophrenia patients:

1. Aged 18 years old or older;
2. Diagnosis of schizophrenia or other psychotic disorder (Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5);
3. Treatment resistance according to the Treatment Response and Resistance in Psychosis (TRRIP) Working Group consensus criteria. This requires a PANSS score of more than 70 and the presence of at least one positive and one negative symptom rated as ≥ 4 on the Positive and Negative Syndrome Scale (PANSS) and at least moderate functional impairment on the Social and Occupational Function Assessment Scale (SOFAS) despite at least 2 adequate trials of different antipsychotics;
4. On a stable dose of antipsychotic (no dose changes in the past 1 month);
5. Able to give fully informed written consent and likely to comply with the requirements of the study, after reading the information and consent form, and after having the opportunity to discuss the study with the investigator or his delegate;
6. Capacity to provide informed consent, as judged by an investigator and as assessed by the McArthur scale;
7. Ability to communicate satisfactorily with the investigator and to participate in, and comply with the requirements of the entire study.

Exclusion criteria for treatment-resistant schizophrenia patients:

1. History of significant co-morbid central nervous system (CNS) disorder (including significant head trauma or significant loss of consciousness, Parkinson's Disease, Epilepsy, Alzheimer's Dementia, Huntington's Disease);
2. Current use of medication with recognized effect on glutamatergic signaling (e.g. lamotrigine, lithium, carbamazepine, opiates, and psychostimulants) OR medication that is known to interact with riluzole (eg: ciprofloxacin, combined hormonal contraceptives, enoxacin, fluvoxamine, charcoal boiled (grilled) foods, methoxasalen, rucaparib, osilodrostat, mexiletine, nicergoline, pipemidic acid, rifampicin, tiabendazole, vemurafenib);
3. Any absolute contra-indication to riluzole according to the British National Formulary (such as interstitial lung disease, current pregnancy or lactation, severe hepatic impairment liver function tests more than 3x Upper limit of normal, acute porphyria, pancreatitis);
4. Pregnancy and/or breast-feeding;
5. Substance dependence/abuse other than to cigarettes;
6. Current high suicide risk or other significant safety risk as judged by the patient's psychiatrist or study physician;
7. Current homicidal ideation or intent;
8. Participation in a clinical study of unlicensed medicines within the previous 30 days;
9. Clinically relevant abnormal findings at the screening assessment as judged significant by the principal investigator (e.g.: history of liver disease or transaminases more than 2 times the upper limit of normal);
10. Presence of other acute or chronic illness or history of chronic illness sufficient to invalidate the volunteer's participation in the study or raise safety concerns;
11. Any risk factors for liver damage (eg. alcohol dependence or history of liver disease) or patients who are receiving potentially hepatotoxic medications;
12. Likelihood that the subject will not comply with study requirements or other reason the investigator judges the subject is not suitable;
13. Objection by subject's physician;
14. Any contraindication to MRI scanning (e.g. metallic implants);
15. Any comorbidity that could compromise scanning safety (e.g. severe asthma).

Inclusion criteria for treatment-responsive schizophrenia patients:

1. Aged 18 years old or older;
2. Diagnosis of schizophrenia or other psychotic disorder (Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5);
3. On a stable dose of antipsychotic (no dose changes in the past 1 month);
4. Able to give fully informed written consent and likely to comply with the requirements of the study, after reading the information and consent form, and after having the opportunity to discuss the study with the investigator or his delegate;
5. Capacity to provide informed consent, as judged by an investigator and as assessed by the McArthur scale;
6. Ability to communicate satisfactorily with the investigator and to participate in, and comply with the requirements of the entire study.

Exclusion criteria for treatment-responsive schizophrenia patients:

1. Treatment resistance according to the Treatment Response and Resistance in Psychosis (TRRIP) Working Group consensus criteria;
2. History of significant co-morbid CNS disorder (including significant head trauma or significant loss of consciousness, Parkinson's Disease, Epilepsy, Alzheimer's Dementia, Huntington's Disease);
3. Substance dependence/abuse other than to cigarettes;
4. Current high suicide risk or other significant safety risk as judged by the patient's psychiatrist or study physician;
5. Current homicidal ideation or intent;
6. Participation in a clinical study of unlicensed medicines within the previous 30 days;
7. Likelihood that the subject will not comply with study requirements or other reason the investigator judges the subject is not suitable;
8. Objection by subject's physician;
9. Any contraindication to MRI scanning (e.g. metallic implants);
10. Any comorbidity that could compromise scanning safety (e.g. severe asthma);

Inclusion criteria for healthy controls:

1. Aged 18 years old or older;
2. No diagnosis of schizophrenia, schizophreniform or any psychotic disorder;
3. Sufficient understanding of the nature of the study and any hazards of participating in it;
4. Ability to communicate satisfactorily with the investigator and to participate in, and comply with the requirements of the entire study;
5. Willingness to give written consent to participate after reading the information and consent form, and after having the opportunity to discuss the study with the investigator or his delegate;
6. Capacity to provide informed consent, as judged by an investigator.

Exclusion criteria for healthy controls

1. Co-morbid psychiatric or other CNS disorder;
2. Family history of Schizophrenia or Psychotic disorders;
3. History of head trauma or loss of consciousness;
4. Substance dependence/abuse other than to cigarettes;
5. Presence of acute or chronic illness or history of chronic illness sufficient to invalidate the volunteer's participation in the study or make it unnecessarily hazardous and judge significant by the principal investigator;
6. Likelihood that the volunteer will not comply with the requirements of the study or other reason the investigator judges the subject is not suitable;
7. Objection by a General Practitioner (GP), or another doctor responsible for their treatment, to the healthy control entering study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in glutamate levels (using magnetic resonance spectroscopy) pre- and post-riluzole administration | Brain measurements will be conducted at baseline (day -7 to day -1 before riluzole administration), day 7 and day 56 (+- 14 days)
  Change in glutamate levels will be assessed (using magnetic resonance spectroscopy) in treatment-resistant schizophrenia patients compared with controls and patients without treatment-resistant schizophrenia

SECONDARY OUTCOMES:
Correlation of glutamate (using magnetic resonance spectroscopy) with brain functional measures at baseline (using functional magnetic resonance imaging) | Brain measurements will be conducted at baseline (day -7 to day -1 before riluzole administration), day 7 and day 56 (+- 14 days)
Longitudinal change in glutamate levels (using magnetic resonance spectroscopy) correlated with longitudinal change in brain functional measures (using functional magnetic resonance imaging) | Brain measurements will be conducted at baseline (day -7 to day -1 before riluzole administration), day 7 and day 56 (+- 14 days)
Longitudinal change in glutamate levels (using magnetic resonance spectroscopy) correlated with changes in psychopathology | Brain measurements will be conducted at baseline (day -7 to day -1 before riluzole administration), day 7 and day 56 (+- 14 days)
  Changes in psychopathology assessed using rating scales Positive and Negative Syndrome Scale (PANSS), Clinical Global Impression scale (CGI), Calgary Depression Scale for Schizophrenia (CDSS), Montgomery and Asberg Depression Rating Scale (MADRS), Hopkins Verbal Learning Test (HVLT) and a computerised cognitive task

CONTACTS AND LOCATIONS:
Overall Officials: Oliver D Howes, Principal Investigator — King's College London
Locations (1):
- Institute of Psychiatry, Psychology and Neuroscience, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No